CLINICAL TRIAL: NCT05449652
Title: Are Exercise Prescriptions for Patients With Cardiovascular Disease, Made by Physiotherapists, in Agreement With International Guidelines?
Brief Title: Exercise Prescriptions for Patients With Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Dominique Hansen, Professor, Hasselt University
Other Study IDs: AXXON
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Cardiovascular Diseases
Keywords: physiotherapy; exercise prescription; cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: To prescribe exercise prescription for CVD patients — To prescribe exercise intensity, frequency, session duration, program duration, and exercise type (endurance or strength training) for the same three patient cases

SUMMARY:
Physiotherapists are often confronted with patients with (elevated risk for) cardiovascular disease (CVD), even when this is not the primary indication for physiotherapy. Hence, physiotherapists should be able to provide evidence-based exercise advice to these patients, but this has not been assessed. The aim of this study was therefore to assess whether exercise prescriptions by physiotherapists to patients with CVD are in accordance with international recommendations.

DETAILED DESCRIPTION:
In this prospective observational survey, forty-seven Belgian physiotherapists agreed to prescribe exercise intensity, frequency, session duration, program duration, and exercise type (endurance or strength training) for the same three patient cases. Exercise prescriptions were compared between clinicians and relations with clinician characteristics were studied. In addition, the agreement between physiotherapists' exercise prescriptions and those from international recommendations (based on a maximal score of 60/per case) was assessed.

ELIGIBILITY:
Inclusion Criteria: Currently professionally active Flemish physiotherapists

Exclusion Criteria: Not having access to a device that allows the use of the EXercise Prescription in Everyday practice & Rehabilitative Training (EXPERT) tool.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Professionaly active Flemish physiotherapists.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Exercise intensity | February - April 2022
  Assessment of the prescription of exercise intensity (expressed in heart rate in beats per minute)
Exercise frequency | February - April 2022
  Assessment of exercise frequency (expressed in number of exercise sessions per week)
Session duration | February - April 2022
  Assessment of session duration (expressed in number of minutes)
Program duration | February - April 2022
  Assessment of program duration (expressed in number of weeks)
Exercise type | February - April 2022
  Aerobic exercise or strength exercise
Total exercise volume | February - April 2022
  Multiplication of number of prescribed weeks, number of prescribed sessions/week, prescribed individual session duration and prescribed exercise intensity

SECONDARY OUTCOMES:
Association between exercise prescriptions and clinician characteristics' | February - April 2022
  Relations between exercise prescriptions (intensity, frequency, session/program duration, exercise type) and clinician characteristics (age, gender, education, experience,...) were studied.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Hansen, Prof, Principal Investigator — Hasselt University
Locations (1):
- Hasselt University, Diepenbeek, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marinus N, Cornelissen V, Meesen R, Coninx K, Hansen D. Are exercise prescriptions for patients with cardiovascular disease, made by physiotherapists, in agreement with European recommendations? Eur J Cardiovasc Nurs. 2024 Apr 12;23(3):230-240. doi: 10.1093/eurjcn/zvad065. PMID 37439451